CLINICAL TRIAL: NCT05925829
Title: Stromal Vascular Fraction and Autologous Activated Platelet-Rich Plasma Combination in Treatment of Type 2 Diabetes
Brief Title: Stromal Vascular Fraction and Autologous Activated Platelet-Rich Plasma Combination in Treating Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hayandra Peduli Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YHP005/Riset/2023
Record Dates: First submitted 2023-06-09; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2; Platelet-rich Plasma; Stromal Vascular Fraction
Keywords: glycosylated hemoglobin A1c; platelet-rich plasma; stromal vascular fraction; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (1):
- SVF and aaPRP treatment (Experimental): Patients treated with SVF and aaPRP
  Interventions: Biological: SVF and aaPRP

INTERVENTIONS:
Biological: SVF and aaPRP — Stromal vascular fraction and autologous activated platelet-rich plasma

SUMMARY:
This study was a retrospective study on type 2 diabetes patients that were treated with autologous stromal vascular fraction (SVF) and autologous activated platelet-rich plasma (aaPRP) measuring HbA1c level at baseline, 1-month, 3-month, 6-month, and 12-month post-treatment.

DETAILED DESCRIPTION:
The preparation of SVF used the H-Remedy (Jakarta, Indonesia) method invented by HayandraLab. Manual liposuction was performed to collect the lipoaspirate. The aaPRP was prepared using an in-house method of HayandraLab. The SVF pellet was resuspended in 0.9% normal saline, resulting in a total of 22 mL SVF suspension. 7 mL of cell suspension was used for quality control. A total of 15 mL SVF suspension was mixed with 3 mL aaPRP. A total of 20 mL of SVF and aaPRP suspension was injected into an infusion bag which contained 250 ml of 0.9% normal saline. The mixture of SVF and aaPRP was then infused intravenously to each patient for a duration of around 30 minutes. The infusion was given on the day of the patient's lipoaspiration procedure. The patients underwent three subsequent infusions of SVF and aaPRP combination, followed by four aaPRP infusions. These therapy sessions were scheduled with a 2-weeks interval.

Inclusion criteria:

1. Patients who were diagnosed with type 2 diabetes (T2D) for at least 2 years with the diagnosis of T2D and treatment with oral anti-hyperglycemic therapy with metformin were in accordance with the guideline for management and prevention of T2D by the Indonesian Society of Endocrinology.
2. Patients who have undergone standard oral anti-hyperglycemic therapy with metformin and had not been able to reach normal HbA1c level with the medication
3. Patients who underwent autologous SVF-aaPRP therapy between January until December 2017

Exclusion criteria

1. Patients who were pregnant
2. Patients who were below 18 years of age
3. Patients who were on insulin therapy

ELIGIBILITY:
Inclusion Criteria:

* patients who were diagnosed with T2D for at least 2 years
* patients who have undergone standard oral anti-hyperglycemic therapy with metformin and had not been able to reach normal HbA1c level with the medication
* patients who underwent autologous SVF-aaPRP therapy between January until December 2017

Exclusion Criteria:

* patients who were pregnant
* patients who were below 18 years of age
* patients who were on insulin therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of SVF and aaPRP in Type 2 Diabetes Patients | Change of baseline HbA1c level at 1 month, 3 months, 6 months, and 12 months
  HbA1c level at baseline, 1-month, 3-month, 6-month, and 12-month post-treatment
Safety of SVF and aaPRP in Type 2 Diabetes Patients | Up to 12 months
  Adverse events related with SVF and aaPRP treatment such as hematoma, infection, profuse bleeding, vessel puncture, intravascular administration of the cell preparation with potential phlebitis and/or distal embolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Hayandra Peduli Foundation, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No
HbA1c level at baseline, 1-month, 3-month, 6-month, and 12-month post-treatment Adverse events post-treatment